CLINICAL TRIAL: NCT02898701
Title: Does Practice Beyond Performance Plateau Improve Motor Learning in Healthy Adults?
Brief Title: Does Overpractice Improve Motor Learning?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Genevieve Olivier, PhD Student, Physical Therapist, Teaching Assistant, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB_00085515
Record Dates: First submitted 2016-09-07; First posted 2016-09-13 (Estimated); Last update posted 2021-06-15 (Actual); Status verified 2021-06

CONDITIONS: Aging
Keywords: Motor Learning; Dose of Motor Practice; Postural Control; Serial Reaction Time Task; Retention; Transfer; Overpractice; Overtraining; Overlearning

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No Overpractice (NoOVP) (Active Comparator): Subjects will perform the intervention (i.e., motor practice of a standing serial reaction time task) according to the practice schedule until they reach a performance plateau on the repeated sequence. At that time, members of the NoOVP group will cease practicing.
  Interventions: Behavioral: Motor Practice of a Standing Serial Reaction Time Task
- Overpractice (OVP) (Experimental): Subjects will perform the intervention (i.e., motor practice of a standing serial reaction time task) according to the practice schedule until they reach a performance plateau on the repeated sequence. At that time, members of the OVP group will continue to practice as part of the overpractice phase until they have completed 100% overpractice.
  Interventions: Behavioral: Motor Practice of a Standing Serial Reaction Time Task
- Standard of Care (SoC) (Active Comparator): Subjects will perform the intervention (i.e., motor practice of a standing serial reaction time task) until they have performed 144 practice trials over the course of one day. At that time, members of the SoC group will cease practicing.
  Interventions: Behavioral: Motor Practice of a Standing Serial Reaction Time Task

INTERVENTIONS:
Behavioral: Motor Practice of a Standing Serial Reaction Time Task — Subjects will perform a standing serial reaction time task on a step reaction mat. Subjects will step to a series of targets, based on a series of stimuli that are presented. One trial is composed of two 12-step sequences. One of the 12-step sequences is random, while the other is a repeated sequence; sequences are presented in random order. After each trial, the subject rests for 25 seconds. Six trials equal 1 block of practice, which is followed by a 4 minute rest break. After each block, feedback is provided about average response time (RT) on all steps included in the block. One complete day of practice consists of 6 blocks of practice in which each block consists of 6 trials.

SUMMARY:
This study contains two pilot studies: 1) one study will investigate practice dosage of a postural stepping task in healthy young individuals in order to determine an operational definition of performance plateau, and 2) the other study will investigate whether practicing beyond reaching a performance plateau improves learning of a postural stepping task in healthy older adults, compared to discontinuing practice immediately after reaching a performance plateau. The investigators hypothesize that the group that continues to practice beyond reaching their performance plateau will learn and retain the motor task better than the other group.

DETAILED DESCRIPTION:
What is the ideal amount, or dose, of practice needed for a person to learn a motor skill? Studies suggest that "more is better," but the optimal dose of motor practice is unknown. Motor learning is defined as a set of internal processes leading to a relatively permanent change in the capability for a motor skill. Older adults and people with neurological disorders have a critical need to learn and relearn motor skills to remain independent, but standard clinical rehabilitation currently provides practice doses that are insufficient to result in motor learning. Under-dosing of practice results in sub-optimal clinical outcomes, while research studies that are dosed insufficiently to identify between-group differences are prone to misinterpretation. Therefore, it is essential for both clinical care and for research that we determine the practice dose needed to optimize motor learning.

Performance curves (i.e., plots of the average performance of a group or individual for each of a number of practice trials or blocks of trials) demonstrate that performance improves (e.g., error decreases or speed increases) during practice, until a point at which performance improvement begins to plateau. Additional practice provided beyond the point at which an individual reaches a performance plateau will be termed overpractice. Amounts of practice that are insufficient to reach a plateau tend not to demonstrate motor learning, while overpractice typically results in retention of the practiced task.

Pilot Study #1: The first pilot study will include healthy young adults who are randomly assigned to practice a postural stepping task for one day, or for five consecutive days of practice. The investigators will use this data to determine an operational definition (i.e., a mathematical definition) of performance plateau. This definition will be used to differentiate the groups in Pilot Study #2.

Pilot Study #2: The second pilot study will include healthy older adults who will be divided into three groups: a standard of care group (i.e. very low dose), an overpractice group, and a no overpractice group. All groups will practice a postural stepping task. The experimental group will be the overpractice (OVP) group, in which each participant will complete 100% additional practice trials after reaching their performance plateau. In contrast, the two active control groups will be the no overpractice (NoOVP) group (in which each participant will stop practicing immediately after reaching a performance plateau), and the standard of care (SoC) group (in which each participant will perform one block of practice).

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for individuals considered healthy older adults will be: (a) 60-95 years of age.
* Inclusion criteria for individuals considered healthy young adults will be: (a) 18-45 years of age.

Exclusion Criteria will include the following for all individuals:

* acute medical problems
* uncorrected vision loss
* any other conditions that affect their mobility or balance which might affect their ability to perform the motor task (arthritis, orthopedic complications, metabolic, vestibular, etc)
* Montreal Cognitive Assessment score <26
* non-english speaking

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2020-03-17 (Actual)

PRIMARY OUTCOMES:
Retention on the Postural Stepping Task | 3 or 4 days after training ends (i.e., 2 or 3 days of no training prior to retention test)
  Retention is the ability to maintain performance improvements of a motor skill after a period of no practice. Response time (RT) is collected & defined as reaction time (amount of time from stimulus presentation to initial release of foot from electrode) plus movement time (amount of time from initial release of foot to foot reaching target). The first half of Block 1 of Day 1 serves as the pre-test performance. The primary outcome measure is the difference in the RT between pre-test and retention test. A decrease in RT over the course of practice reflects an increased response speed and a corresponding improvement in performance.

SECONDARY OUTCOMES:
Transfer to an Untrained Task | 3 or 4 days after training ends (i.e., 2 or 3 days of no training prior to retention test)
  Transfer is the gain or the loss of proficiency on one task as a result of previous practice or experience on another task. The secondary outcome measure is improvement on the transfer task. The transfer task is the 4 Square Step Test, and is scored based on the number of seconds the participant requires to complete the test. Each participant will perform the 4 Square Step Test at baseline (pre-test) and will perform it three days after the acquisition phase ends (post-test). The post-test score will be subtracted from pre-test score, which will provide a transfer test change score. A positive number will suggest improvement, while a negative number will suggest that the participants worsened on the transfer task.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Trewartha KM, Garcia A, Wolpert DM, Flanagan JR. Fast but fleeting: adaptive motor learning processes associated with aging and cognitive decline. J Neurosci. 2014 Oct 1;34(40):13411-21. doi: 10.1523/JNEUROSCI.1489-14.2014. PMID 25274819
- [Background] Clark BC, Manini TM. Functional consequences of sarcopenia and dynapenia in the elderly. Curr Opin Clin Nutr Metab Care. 2010 May;13(3):271-6. doi: 10.1097/MCO.0b013e328337819e. PMID 20154609
- [Background] Kleim JA, Jones TA. Principles of experience-dependent neural plasticity: implications for rehabilitation after brain damage. J Speech Lang Hear Res. 2008 Feb;51(1):S225-39. doi: 10.1044/1092-4388(2008/018). PMID 18230848
- [Background] Lang CE, Macdonald JR, Reisman DS, Boyd L, Jacobson Kimberley T, Schindler-Ivens SM, Hornby TG, Ross SA, Scheets PL. Observation of amounts of movement practice provided during stroke rehabilitation. Arch Phys Med Rehabil. 2009 Oct;90(10):1692-8. doi: 10.1016/j.apmr.2009.04.005. PMID 19801058
- [Background] Lohse KR, Lang CE, Boyd LA. Is more better? Using metadata to explore dose-response relationships in stroke rehabilitation. Stroke. 2014 Jul;45(7):2053-8. doi: 10.1161/STROKEAHA.114.004695. Epub 2014 May 27. PMID 24867924
- [Background] Lang CE, MacDonald JR, Gnip C. Counting repetitions: an observational study of outpatient therapy for people with hemiparesis post-stroke. J Neurol Phys Ther. 2007 Mar;31(1):3-10. doi: 10.1097/01.npt.0000260568.31746.34. PMID 17419883
- [Background] Krueger WFC. Further studies in overlearning. Journal of Experimental Psychology. 1930;13(2):152-163.
- [Background] Melnick MJ. Effects of overlearning on the retention of a gross motor skill. Res Q. 1971 Mar;42(1):60-9. No abstract available. PMID 5279070
- [Background] Schendel JD, Hagman JD. On sustaining procedural skills over a prolonged retention interval. Journal of Applied Psychology. 1982;67(5):605-610.
- [Background] Driskell JE, Willis RP, Copper C. Effect of overlearning on retention. Journal of Applied Psychology. 1992;77(5):615-622.
- [Background] Jones MB. Nonimposed overpractice and skill retention. DTIC Document;1986.
- [Derived] Olivier GN, Dibble LE, Paul SS, Lohse KR, Walter CS, Marker RJ, Hayes HA, Foreman KB, Duff K, Schaefer SY. Personalized practice dosages may improve motor learning in older adults compared to "standard of care" practice dosages: A randomized controlled trial. Front Rehabil Sci. 2022 Aug 3;3:897997. doi: 10.3389/fresc.2022.897997. eCollection 2022. PMID 36189036